CLINICAL TRIAL: NCT05095090
Title: Observational Cohort Study of Hospitalised Patients With Acute Respiratory Conditions
Brief Title: Study of Hospitalised Patients With Acute Respiratory Conditions
Acronym: CHESTY
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Leicester (Other)
Collaborators: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0822
Record Dates: First submitted 2021-09-08; First posted 2021-10-27 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Acute Respiratory Disease; COPD Exacerbation Acute; Asthma; Pneumonia
Keywords: Asthma; COPD (Chronic Obstructive Pulmonary Disease); Pneumonia; ILD (Interstitial Lung Diseases); Pulmonary Embolism; Pleural Diseases; Bronchiectasis
MeSH Terms: conditions — Asthma; Pneumonia; Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial; Pulmonary Embolism; Pleural Diseases; Bronchiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — As part of the optional blood tests specified above, specific samples can be analysed for genetic testing related to respiratory conditions. The participants will decide when signing the consent form, if they are happy for their samples to undergo genetic analysis. The results will not be communicated back to the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hospitalised Patients: Participants admitted to hospital with an acute respiratory condition including exacerbation of an underlying physician diagnosed chronic lung disease.
- Matched Controls: The study will include matched controls (non-hospitalised patients with stable chronic respiratory conditions or healthy volunteers) to compare the exploratory endpoints. The number of the matched controls will not exceed 25% of the main study recruitment.

SUMMARY:
This observational study aim to characterise patients admitted to hospital with an acute respiratory condition, or acute worsening of their chronic lung condition. This will enable identification of predictors of future risk, as well as develop potential interventions targets.

DETAILED DESCRIPTION:
This will be an observational cohort study, recruiting patients who have been admitted to hospital with an acute respiratory condition. This can include exacerbation of an existing chronic lung disease such as asthma, COPD, interstitial lung disease, bronchiectasis and pleural disease, or contracting an acute illness including pulmonary embolism, pneumonia, or any other respiratory infection. The patients will be screened and recruited whilst still hospitalised and followed up for one year after discharge. The participants will undergo a baseline study visit while in hospital, with the option to have further follow up visits (up to three occasions) in the following year to assess clinical recovery.

The participants will be offered the choice to undertake the follow up assessments via any of the following routes:

* a telephone consultation or
* a face to face visit either in the Biomedical Research Centre (BRC) or
* during a research visit from another ethically approved study or
* during routine clinical follow up organised by the hospital clinical team.

The participants can choose not to attend any further follow up visits after discharge. Any planned clinical follow-up arranged by the hospital team will occur according to clinical needs. If the participant is re-admitted during the 12 months after enrolment, assessments identical to the baseline visit can be repeated.

A final remote visit will be carried out at 12 months post-discharge (+/- 1 month) to collect data about health care utilisation (e.g. hospitalisation rate, length of stay in hospital, death rate, antibiotic/steroid prescriptions) from both primary and secondary healthcare records. The participants are not required to attend this final visit as data will be collected remotely.

ELIGIBILITY:
Hospitalised Patients

Inclusion Criteria:

1. Hospital admission with an acute respiratory diagnosis
2. Participant is willing & able to give informed consent for participation in the study
3. Aged 18 years or above
4. Able (in the Investigators opinion) & willing to comply with all study requirements

Exclusion Criteria:

1. Unstable or life-threatening cardiac disease including myocardial infarction or unstable angina during current admission.
2. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
3. Known pregnancy

Matched Controls

Inclusion Criteria:

1. Aged 18 years or above
2. Patients with stable chronic respiratory conditions or healthy volunteers
3. Able (in the Investigators opinion) & willing to comply with all study requirements

7.3.2 Exclusion Criteria:

1. Hospitalised due to an acute respiratory illness in the last 6 weeks prior to consent
2. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
3. Known pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants admitted to hospital with an acute respiratory condition including exacerbation of an underlying physician diagnosed chronic lung disease. The study will include matched controls (non-hospitalised patients with stable chronic respiratory conditions or healthy volunteers). Co-participation in other ethically approved studies including interventional trials is permissible.
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
30 days hospital re-admission rate | 30 days
  To calculate the percentage of readmission due to the same acute respiratory illness within 30 days from consent
Length of index hospital admission stay | Variable (up to 52 weeks)
  To calculate the length of the index hospital stay
30 days mortality rate | 30 days
  To calculate the percentage of mortality within 30 days from consent

SECONDARY OUTCOMES:
Total number of hospital readmission due to same underlying chronic lung disease. | 52 weeks
  To evaluate the number of hospital readmission episodes due to same underlying chronic lung disease over a 52 weeks period.
Total number of non-hospitalised exacerbations of underlying chronic lung disease | 52 weeks
  To evaluate the number of non-hospitalised exacerbations of chronic lung disease e.g. asthma, Chronic Obstructive Pulmonary Diseases (COPD), etc. over 52 weeks
Time from consent to death (respiratory causes and all causes) | 52 weeks
  To measure the time from consent to death within 52 weeks from consent. This will include both respiratory and all causes of mortality

OTHER OUTCOMES:
Assessment of breathlessness using eMRC dyspnoea scale | 52 weeks
  To evaluate the degree of breathlessness at baseline and following recovery from acute respiratory illness using Extended MRC dyspnoea scale(eMRC). eMRC dyspnoea scale ranges from 1 to 5b with higher score indicates worse outcomes.
Assessment of quality of Life/symptoms using St. George's Respiratory Questionnaire (SGRQ) | 52 weeks
  St. George's Respiratory Questionnaire (SGRQ) is a disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. Scores range from 0 to 100, with higher scores indicating more limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Greening, PhD, MRCP, Principal Investigator — NIHR Respiratory Biomedical Research Centre, Leicester
Locations (1):
- Glenfield Hospital, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No